CLINICAL TRIAL: NCT03366454
Title: Implementing a Combination of Clinical Parameters (Rapid Diagnostic Tests (RDTs), Biomarkers, and Standard of Care Procedures (SoCs) for the Etiology Diagnoses of Pneumonia in Pediatric Patients to Improve Clinical Management in Indonesia.
Brief Title: Implementing a Combination of Clinical Parameters, Biomarkers and SoCs for the Etiology Diagnoses of Pneumonia in Pediatric Patients
Acronym: PEER-PePPes
Status: Completed | Type: Observational
Sponsor: INA-RESPOND Secretariat (Other)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency); Indonesia Research Partnership on Infectious Disease (INA-RESPOND) (Unknown)
Responsible Party: Sponsor-Investigator, INA-RESPOND Secretariat, dr. Herman Kosasih, PhD, Ina-Respond
Organization: Ina-Respond (Other)
Other Study IDs: INA201; U1111-1263-2368 (Other: WHO UTN Number)
Record Dates: First submitted 2017-11-08; First posted 2017-12-08 (Actual); Results first posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Pneumonia
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Subjects must be willing to allow storage of left over specimens (whole blood, serum, urine, NPS, sputum/induced sputum) and isolate from culture (if available)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Participants who meet the inclusion and exclusion criteria will be enrolled and then having a daily follow up for maximum of 13 days' hospitalization. Next follow up will be taken time at day 14th after hospitalization date, either on ward or policlinic. The participations will be ended by day 30th after hospitalization date when the called follow up is done by investigator.

DETAILED DESCRIPTION:
This study will collect demographic data, medical history, clinical data, treatment, and risk factors of pneumonia. The study also record the supporting examination results include but not limited to Complete Blood Count (CBC) results, blood gas analyses result, CRP, PCT, culture result, rapid test for influenza, Respiratory Syncytial Virus (RSV), legionella, and chest X-ray. In order to produce a robust data, this study will conduct the serological and molecular tests at the reference laboratory.

Whole blood, serum, urine, Nasal Pharyngeal Swab (NPS), sputum/induced sputum, and other respiratory specimens (if available) will be collected for storage and testing at enrollment. Plasma from 48-72 hours after hospitalization and left-over respiratory specimens on day 2 and 3 of hospitalization will also be collected to be stored. For additional, at day 14th after hospitalization serum will be processed from 4 mL of blood for archiving and testing at the reference laboratory.

This study will be conducted at following INA-RESPOND sites:

* RSU Kabupaten Tangerang, Tangerang
* RSUP Dr. Kariadi, Semarang
* RSUP Dr. Sardjito, Yogyakarta RSU Kabupaten Tangerang located in Banten province is type B or district referral hospital. While RSUP Dr Kariadi in Semarang and RSUP Dr Sardjito in Yogyakarta are type A hospital which is a level of province referral. Maximum duration for participants' accrual will be 2 years since the first participant enrolled. However, the study laboratory testing may take up to 6 months to be completed.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric inpatients whose ages range from 2 months to 5 years
* Meet the case definition for pneumonia which is cough or fever with at least one other following symptoms:

  * Shortness of breath
  * Tachypnea
  * Grunting
  * Crackles/rhonchi
  * Decreased vesicular breath sound
  * Bronchial breath sound
  * Chest x-ray consistent with pneumonia
* Comply with all study procedures including to store required specimens for diagnostic testing and archiving.

Exclusion Criteria:

* Being Hospitalized for more than 24 hours at enrollment
* Having a cancer or history of cancer
* Having a history of long term exposed of steroid (at the minimum of 2 months)
* Having any condition that might interfere with study procedure and compliance (based on clinicians' judgement)

Ages: 2 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Hospitalized patients with pneumonia whose ages range from 2 months to 5 years. This is a preliminary study to characterize the pathogens present in this cohort. The number of participants' that will be enrolled is based on the number of pneumonia cases in 5 years old children or less, which is approximately 100 patients per year in each hospital. Estimating that 50% of them failed to satisfy the inclusion and exclusion criteria, this study plan to enroll 50 participants per site per year, or a total of 275 participants.
Sampling Method: Non-Probability Sample
Enrollment: 188 (Actual)
Dates: Start 2017-07-04 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Herman Kosasih, PhD, Principal Investigator — Ina-Respond
Locations (4):
- Indonesia (4):
  - University of Diponegoro/ Dr. Kariadi Hospital, Semarang, Central Java
  - University of Gadjah Mada/ Dr. Sardjito Hospital, Yogyakarta, DIY Yogyakarta
  - RSU Kabupaten Tangerang, Tangerang, West Java
  - An-Nisa Hospital, Tangerang, West Java

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lokida D, Farida H, Triasih R, Mardian Y, Kosasih H, Naysilla AM, Budiman A, Hayuningsih C, Anam MS, Wastoro D, Mujahidah M, Dipayana S, Setyati A, Aman AT, Lukman N, Karyana M, Kline A, Neal A, Lau CY, Lane C. Epidemiology of community-acquired pneumonia among hospitalised children in Indonesia: a multicentre, prospective study. BMJ Open. 2022 Jun 21;12(6):e057957. doi: 10.1136/bmjopen-2021-057957. PMID 35728910

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period was done from July 2017 to September 2019
Pre-assignment Details: From total target 275 subjects only achieved 188 subjects enrolled
Groups:
- Hospitalized Pediatric Participants With Pneumonia: Hospitalized pediatric patients with pneumonia at acute episode.
Period: Overall Study
Arm/Group | Hospitalized Pediatric Participants With Pneumonia
Started | 188
Completed | 188
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Hospitalized Pediatric Participants With Pneumonia
Number analyzed (Participants) | 188
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 188
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Median (Inter-Quartile Range); unit: months] | 9 [5 to 20]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 85
  Male | 103
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 188
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 188
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Indonesia | 188

OUTCOME MEASURES:

1. Primary Outcome: White Blood Cells and Absolute Neutrophil Count Cut-off Levels for Distinguishing of Viral and Bacterial/Mixed Pathogens
Description: The area under the receiver operating curve (AUROC) for WBC and ANC count at enrolment was used to characterize their utility for discriminating bacterial/mixed and viral pathogens and for determining the best cut-off values. For this analysis, a total of 155 subjects with confirmed bacterial/mixed or viral infections were included.
Time Frame: Total length of time the subject will be in the study is one month after enrollment.
Population: All subjects with confirmed etiology.
Measure: Number; unit: 10^3 cells/microliter
Groups:
- White Blood Cells Count Cut-off Levels for Distinguishing of Viral and Bacterial/Mixed Pathogens: The WBC count data at enrolment was used to characterize their utility for discriminating bacterial/mixed and viral pathogens and for determining the best cut-off values. For this analysis, a total of 155 subjects with confirmed bacterial/mixed or viral infections were included.
- Absolute Neutrophil Count Cut-off Levels for Distinguishing of Viral and Bacterial/Mixed Pathogens: The ANC count data at enrolment was used to characterize their utility for discriminating bacterial/mixed and viral pathogens and for determining the best cut-off values. For this analysis, a total of 155 subjects with confirmed bacterial/mixed or viral infections were included.
Arm/Group | White Blood Cells Count Cut-off Levels for Distinguishing of Viral and Bacterial/Mixed Pathogens | Absolute Neutrophil Count Cut-off Levels for Distinguishing of Viral and Bacterial/Mixed Pathogens
Number analyzed (Participants) | 155 | 155
10^3 cells/microliter | 12.2 | 6.15
Statistical Analysis 1: Comparison: White Blood Cells Count Cut-off Levels for Distinguishing of Viral and Bacterial/Mixed Pathogens; ROC curve analysis was performed to evaluate outcome. The Area Under the Curve (AUC) was calculated along with a 95% confidence interval and statistical significance (p-value); Test type: Other; p = 0.0048, ROC Curve Analysis; AUC = 0.6692, 95% CI 2-sided [0.5649 to 0.7735], Standard Error of Mean 0.05322
Statistical Analysis 2: Comparison: Absolute Neutrophil Count Cut-off Levels for Distinguishing of Viral and Bacterial/Mixed Pathogens; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.0029, ROC Curve Analysis; AUC = 0.6892, 95% CI 2-sided [0.5870 to 0.7914], Standard Error of Mean 0.05213

2. Primary Outcome: Neutrophil Lymphocyte Ratio Cut-off for Distinguishing of Viral and Bacterial/Mixed Pathogens
Description: The area under the receiver operating curve (AUROC) for NLR at enrolment was used to characterize their utility for discriminating bacterial/mixed and viral pathogens and for determining the best cut-off values. For this analysis, a total of 155 subjects with confirmed bacterial/mixed or viral infections were included.
Time Frame: Total length of time the subject will be in the study is one month after enrollment.
Population: All subjects with confirmed etiology.
Measure: Number; unit: ratio
Groups:
- Neutrophil Lymphocyte Ratio Cut-off for Distinguishing of Viral and Bacterial/Mixed Pathogens: The area under the receiver operating curve (AUROC) for NLR at enrolment was used to characterize their utility for discriminating bacterial/mixed and viral pathogens and for determining the best cut-off values. For this analysis, a total of 155 subjects with confirmed bacterial/mixed or viral infections were included.
Arm/Group | Neutrophil Lymphocyte Ratio Cut-off for Distinguishing of Viral and Bacterial/Mixed Pathogens
Number analyzed (Participants) | 155
ratio | 1.34
Statistical Analysis 1: Comparison: Neutrophil Lymphocyte Ratio Cut-off for Distinguishing of Viral and Bacterial/Mixed Pathogens; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.0233, ROC Curve Analysis; AUC = 0.6440, 95% CI 2-sided [0.5335 to 0.7544], Standard Error of Mean 0.05635 — The optimal cutoff value for NLR was determined as 1.335 using the Youden Index

3. Primary Outcome: CRP Cut-off for Distinguishing of Viral and Bacterial/Mixed Pathogens
Description: The area under the receiver operating curve (AUROC) for CRP at enrolment was used to characterize their utility for discriminating bacterial/mixed and viral pathogens and for determining the best cut-off values. For this analysis, a total of 155 subjects with confirmed bacterial/mixed or viral infections were included.
Time Frame: Total length of time the subject will be in the study is one month after enrollment.
Population: All subjects with confirmed etiology.
Measure: Number; unit: mg/dL
Groups:
- CRP Cut-off for Distinguishing of Viral and Bacterial/Mixed Pathogens (mg/L): The area under the receiver operating curve (AUROC) for CRP at enrolment was used to characterize their utility for discriminating bacterial/mixed and viral pathogens and for determining the best cut-off values. For this analysis, a total of 155 subjects with confirmed bacterial/mixed or viral infections were included.
Arm/Group | CRP Cut-off for Distinguishing of Viral and Bacterial/Mixed Pathogens (mg/L)
Number analyzed (Participants) | 155
mg/dL | 5.70
Statistical Analysis 1: Comparison: CRP Cut-off for Distinguishing of Viral and Bacterial/Mixed Pathogens (mg/L); [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.0018, ROC Curve Analysis; AUC = 0.6884, 95% CI 2-sided [0.5962 to 0.7807], Standard Error of Mean 0.04709 — The optimal cut-off value for CRP was determined as 5.70 using the Youden Index

4. Primary Outcome: Procalcitonin Cut-off for Distinguishing of Viral and Bacterial/Mixed Pathogens
Description: The area under the receiver operating curve (AUROC) for PCT at enrolment was used to characterize their utility for discriminating bacterial/mixed and viral pathogens and for determining the best cut-off values. For this analysis, a total of 155 subjects with confirmed bacterial/mixed or viral infections were included.
Time Frame: Total length of time the subject will be in the study is one month after enrollment.
Population: All subjects with confirmed etiology.
Measure: Number; unit: ng/mL
Groups:
- Procalcitonin Cut-off for Distinguishing of Viral and Bacterial/Mixed Pathogens (ng/mL): The area under the receiver operating curve (AUROC) for PCT at enrolment was used to characterize their utility for discriminating bacterial/mixed and viral pathogens and for determining the best cut-off values. For this analysis, a total of 155 subjects with confirmed bacterial/mixed or viral infections were included.
Arm/Group | Procalcitonin Cut-off for Distinguishing of Viral and Bacterial/Mixed Pathogens (ng/mL)
Number analyzed (Participants) | 155
ng/mL | 0.141
Statistical Analysis 1: Comparison: Procalcitonin Cut-off for Distinguishing of Viral and Bacterial/Mixed Pathogens (ng/mL); [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.0007, ROC Curve Analysis; AUC = 0.7063, 95% CI 2-sided [0.6111 to 0.8015], Standard Error of Mean 0.04857 — The optimal cutoff value for PCT was determined as 0.141 using the Youden Index

5. Secondary Outcome: The Etiologies of Pneumonia in Children Expressed in Percentages of Enrolled Subjects.
Description: Any pathogens identified as a cause of pneumonia based on laboratory tests such as culture, serology, and molecular assays.
Time Frame: Total length of time the subject will be in the study is one month after enrollment.
Population: All participants who have specimens to be tested
Measure: Count of Participants; unit: Participants
Arm/Group | Hospitalized Pediatric Participants With Pneumonia
Number analyzed (Participants) | 188
Participants
  Bacterial | 48
  Viruses | 31
  Mixed pathogens | 76
  Unidentified pathogens | 33

6. Secondary Outcome: The Clinical Outcome in Pneumonia Pediatric Subjects
Description: Data and specimens were collected at enrollment and 14 days after enrollment. A telephone interview was done on day 30 to assess the clinical outcome. The outcome report was expressed in percentages of enrolled subjects and the proportions of subjects within each category defined by cured and death.
Time Frame: Total length of time the subject will be in the study is one month after enrollment.
Population: All subjects enrolled with clinical data.
Measure: Count of Participants; unit: Participants
Groups:
- Bacterial Pathogens; Viral Pathogens; Mixed Pathogens; Unidentified Pathogens: Identified etiology based on laboratory testing
Arm/Group | Bacterial Pathogens | Viral Pathogens | Mixed Pathogens | Unidentified Pathogens
Number analyzed (Participants) | 48 | 31 | 76 | 33
Participants
  Cured | 41 | 29 | 71 | 28
  Death | 7 | 2 | 5 | 5

7. Secondary Outcome: The Percentage of Sign and Symptom of SoC Procedure
Description: The percentage of sign and symptom of SoC procedure of pneumonia pediatric subjects expressed in percentages of identified pathogens. The proportion of subjects within each category is defined by bacterial or mixed infections and viral infections. We analyzed only 155 subjects with confirmed etiology for this secondary outcome.
Time Frame: Total length of time the subject will be in the study is one month after enrollment.
Population: All subjects with confirmed etiology.
Measure: Count of Participants; unit: Participants
Groups:
- Bacterial or Mixed Infections: Bacterial or mixed pathogens were identified based on laboratory testing as a caused of pneumonia infection
- Viral Infections: Viral pathogens were identified based on laboratory testing as a caused of pneumonia infection
Arm/Group | Bacterial or Mixed Infections | Viral Infections
Number analyzed (Participants) | 124 | 31
Participants
  Cough | 116 | 27
  Shortness of breath | 116 | 28
  Fever | 105 | 22
  Decreased consciousness | 6 | 0
  Inability to drink | 10 | 2
  Diarrhea | 30 | 1
  Vomiting | 9 | 2
  Seizure | 5 | 1
  Tachypnea | 54 | 13
  Intercostal retraction | 112 | 27
  Ronchi | 115 | 25
  Wheezing | 20 | 2
  Nasal Flaring | 49 | 11
  Chest indrawing | 85 | 18
  Head bobbing | 7 | 2
  Skin rash | 6 | 2
  SpO2 <90% | 29 | 6
  Severe/ very severe pneumonia (WHO classification 2014) | 55 | 16
  Chest X-ray Pleural effusion | 3 | 1
  Chest X-ray- Interstitial infiltrate | 93 | 19
  Chest X-ray-Alveolar infiltrate | 86 | 19

8. Secondary Outcome: Performance of Combined Factors in Differentiating Viral and Bacterial Infections
Description: We explored the combination of significant factors/variables in the multivariate analysis for their overall sensitivity and specificity for discriminating bacterial/mixed and viral infection. The combination variables were CRP ≥5.70 mg/L + fever, CRP ≥5.70 mg/L + dry season, and CRP ≥5.70 mg/L + fever + dry season.
  For this analysis, a total of 155 subjects with confirmed bacterial/mixed or viral infections were included.
Time Frame: Total length of time the subject will be in the study is one month after enrollment.
Population: All subjects with confirmed etiology.
Measure: Number; unit: percentage of participants
Groups:
- CRP ≥5.70 mg/L + Fever; CRP ≥5.70 mg/L + Fever + Dry Season: We explored the combination of significant factors/variables in the multivariate analysis for their overall sensitivity and specificity for discriminating bacterial/mixed and viral infection.
  For this analysis, a total of 155 subjects with confirmed bacterial/mixed or viral infections were included.
- CRP ≥5.70 mg/L + Dry Season: We explored the combination of significant factors/variables in the multivariate analysis for their overall sensitivity and specificity for discriminating bacterial/mixed and viral infection.
  For this analysis, a total of 155 subjects with confirmed bacterial/mixed or viral infections were included. s
Arm/Group | CRP ≥5.70 mg/L + Fever | CRP ≥5.70 mg/L + Dry Season | CRP ≥5.70 mg/L + Fever + Dry Season
Number analyzed (Participants) | 155 | 155 | 155
percentage of participants
  Sensitivity | 62.28 | 40.35 | 35.09
  Specificity | 65.52 | 82.76 | 86.21
  PPV | 87.65 | 90.19 | 90.91
  NPV | 30.64 | 26.09 | 25.25

9. Secondary Outcome: Number of Strains of Circulating Respiratory Viruses and Pathogens in Pediatric Pneumonia Subjects
Description: Any pathogens identified as a cause of pneumonia based on laboratory tests such as culture, serology, and molecular assays. We analyzed only 155 subjects with confirmed etiology for this secondary outcome.
Time Frame: Total length of time the subject will be in the study is one month after enrollment.
Population: All subjects with confirmed etiology.
Measure: Number; unit: participants
Groups:
- Identified Pathogens: Any pathogens identified as a cause of pneumonia based on laboratory tests
Arm/Group | Identified Pathogens
Number analyzed (Participants) | 155
participants
  Streptococcus pneumoniae | 29
  Staphylococcus aureus | 20
  Streptococcus mitis | 4
  Streptococcus pyogenes | 1
  Moraxella catarrhalis | 2
  Haemophilus influenzae non type B | 73
  Klebsiella pneumoniae | 43
  Bordetella pertussis | 7
  Escherichia coli | 5
  Pseudomonas aeruginosa | 4
  Acinetobacter baumannii | 3
  Haemophilus influenzae type B | 2
  Neisseria meningitidis | 1
  Chlamydia pneumoniae | 5
  Mycoplasma pneumonia | 5
  Legionella pneumophila | 1
  RSV A | 15
  RSV B | 36
  Influenza | 25
  Influenza A (H1N1) | 7
  Influenza A (H3N2) | 3
  Influenza B | 14
  PIV 1 | 5
  PIV 3 | 11
  PIV 4 | 1
  hMPV | 11
  Rhinovirus | 10
  Enterovirus | 5
  Bocavirus | 3
  hCoV-NL63 | 2

ADVERSE EVENTS:
Time Frame: 2 years, 2 months
Description: Any untoward or unfavorable medical occurrence in a human subject that occurs within 48 hours of a study-related specimen collection that is possibly, probably, or definitely related to the blood draw or induced sputum. Any event outside of this 48 hour window period will not be considered an AE for this study.
Groups:
- Obervational: Hospitalized pediatric participants with pneumonia
Arm/Group | Obervational
All-Cause Mortality (participants affected / at risk) | 19/188
Serious Adverse Events (participants affected / at risk) | 0/188
Other Adverse Events (participants affected / at risk) | 1/188
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Obervational (N=188)
Hematoma (Skin and subcutaneous tissue disorders) | 1 (1) — Hematoma at the site where blood is drawn

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-03-13): https://cdn.clinicaltrials.gov/large-docs/54/NCT03366454/Prot_SAP_ICF_000.pdf